CLINICAL TRIAL: NCT07097064
Title: Evaluation of the Stereotactic MR-guided Adaptive Radiotherapy for Locally Advanced Pancreatic Cancers
Acronym: RAIPANC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROICM 2024-06 RAI
Record Dates: First submitted 2025-07-17; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Locally Advanced Pancreatic Adenocarcinoma
Keywords: Pancreatic Adenocarcinoma; adaptative radiotherapy
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard cohort (Active Comparator): intensity-modulated conformal radiotherapy (IMRT) 50-54 Gy in 25-30 fractions with concomitant Xeloda 800-825 mg/m2 morning and evening 5 days a week (standard of care according to RECORAD and TNCD).
  Interventions: Combination Product: standard radiotherapy with chemotherapy
- Experimental cohort (Experimental): MRI-guided adaptive stereotactic radiotherapy (extreme hypofractionation) (SMART) 50Gy/ 5 fractions without concomitant chemotherapy.
  Interventions: Radiation: MRI-guided adaptive stereotactic radiotherapy (SMART)

INTERVENTIONS:
Combination Product: standard radiotherapy with chemotherapy — intensity-modulated conformal radiotherapy (IMRT) 50-54 Gy in 25-30 fractions with concomitant Xeloda 800-825 mg/m2 morning and evening 5d/7.
  Arms: Standard cohort
Radiation: MRI-guided adaptive stereotactic radiotherapy (SMART) — MRI-guided adaptive stereotactic radiotherapy (SMART) 50 Gy / 5 fractions without concomitant chemotherapy.
  Arms: Experimental cohort

SUMMARY:
Pancreatic cancer is on the rise, and is set to become the 2nd leading cause of cancer deaths by 2030. Its prognosis is very poor, with a 5-year survival rate of just 5.5%. Curative surgery with chemotherapy improves survival, but only 20% of patients are eligible. For locally advanced forms, radiotherapy, notably in the form of MRI-guided adaptive stereotactic radiotherapy (SMART), is showing promising results in terms of survival and local control, but still requires prospective validation.

DETAILED DESCRIPTION:
In 2016, pancreatic cancer became the 3rd leading cause of cancer death worldwide, and could be the 2nd by 2030. Its prognosis remains very unfavorable, with a 5-year overall survival rate of 5.5%, all stages combined. In France, incidence is on the rise, with 14,100 new cases and 11,400 deaths in 2018. The only therapeutic strategy that has shown a significant improvement in survival is curative surgery followed by adjuvant chemotherapy, but only 20% of patients are eligible. The majority of cases are diagnosed at an advanced or unresectable stage.

For locally advanced cancers (LACC), management is not standardized. Two induction chemotherapy regimens have been validated: FOLFIRINOX and GEMBRAX. The role of radiochemotherapy remains debated. The LAP07 study showed no significant benefit of radiochemotherapy on overall survival, although it did improve progression-free survival and locoregional control.

New techniques such as MRI-guided adaptive stereotactic radiotherapy (SMART) enable more targeted and intense delivery of radiation dose, while protecting organs at risk. Retrospective studies have shown a significant improvement in local control (up to 98% at 1 year) and overall survival (up to 23 months) with this method, compared with conventional radiotherapy. However, prospective studies are still needed to confirm the value of SMART in the management of locally advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven pancreatic adenocarcinoma ;
* Age ≥ 18 years ;
* WHO score 0-1 ;
* Locally advanced according to NCCN 1.2015 recommendations;
* Non-metastatic after TAP scan and MRI of the liver ;
* CA 19.9 < 1000 IU/mL ;
* Completion of at least 4 cycles of induction chemotherapy (Folfirinox and/or Gemzar-Abraxane) with a maximum of 8 courses ;
* Women of childbearing potential must have a pregnancy blood test within a maximum of 7 days before starting the study treatment. A negative result must be documented before study treatment is started. Women without reproductive potential are postmenopausal women or women who have undergone permanent sterilisation (e.g. tubal occlusion, hysterectomy, bilateral salpingectomy) ;
* Effective contraception for women of childbearing age ;
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other study procedures ;
* Patient has given informed, written and express consent ;
* Patient affiliated to a French health insurance scheme.

Exclusion Criteria:

* Other concomitant cancer or history of cancer, with the exception of treated cervical cancer in situ, basal or squamous cell skin carcinoma, superficial bladder tumour (Ta, Tis, and T1) or a tumour with a good prognosis treated curatively without chemotherapy and without evidence of disease in the 3 years prior to inclusion ;
* History of radiotherapy with a foreseeable overlap with the radiotherapy treatment under study (history of abdominal irradiation) ;
* Contraindication to MRI and MRI-guided radiotherapy (claustrophobia, presence of metallic elements etc...) ;
* History of chronic inflammatory disease of the colon or rectum ;
* Women who are pregnant, parturient or breastfeeding ;
* Any other serious concomitant and unbalanced disease or disorder that may interfere with the patient's participation in the study and his/her safety during the study (e.g. severe hepatic, renal, pulmonary, metabolic, or psychiatric disorders) ;
* Legal incapacity (patient under curatorship or guardianship) ;
* History of severe and unexpected reactions to treatment containing a fluoropyrimidine ;
* Hypersensitivity to capecitabine, to used excipients or to fluorouracil ;
* Known complete deficiency of dihydropyrimidine dehydrogenase (DPD) ;
* In patients with severe leukopenia, neutropenia or thrombocytopenia ;
* In patients with severe hepatic insufficiency ;
* Patients with severe renal insufficiency (creatinine clearance less than 30 mL/min) ;
* Recent or concomitant treatment with brivudine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2033-09 (Estimated)

PRIMARY OUTCOMES:
Improvement of local control at 1 year by 20% in the experimental cohort compared with the standard cohort. | From enrollment to one year after treatment completion
  Local control rate, assessed by TAP scan according to RECIST 1.1 criteria (Appendix 8) +/- oesogastroduodenal fibroscopy (FOGD) in case of upper digestive symptomatology not explained by CT scan.
  The local control rate is defined as the proportion of patients without local progression, the time to local progression being defined as the time between the start date of radiotherapy and the date of documented local progression. Patients will be censored at date of death if they die of a carcinological outcome other than local recurrence, or of another cause. Patients without local progression will be censored at the date of last follow-up.

SECONDARY OUTCOMES:
Evaluation of Overall Survival | 1 year after enrollment
  Overall survival (OS) at 1 year, with overall survival defined as the time between the date of starting RT treatment and the date of death from any cause ;
Evaluation of progression-free survival | 1 year after enrollment
  Progression-free survival (PFS) at 1 year, progression-free survival defined as the time between the date of starting RT treatment and the date of 1st documented progression or the date of death from any cause ; Progression will be assessed by TAP, or OGD if suspicion of local recurrence not identified on the scanner (same imaging technique for all patients) ;
Evaluation of Metastasis-free survival | 1 year after enrollment
  Metastasis-free survival (MFS) at 1 year, with MFS defined as the time from the start date of RT treatment to the date of first metastatic progression; Metastatic progression will be assessed using CT-scan
Evaluation of severe acute gastrointestinal toxicity | 90 days after the end of radiotherapy
  Rate of intestinal and gastric toxicity grade > 2 during and in the 90 days following the end of radiotherapy, evaluated according to the CTCAE v5.0 classification
Evaluation of safety (acute and late toxicities of RT) | Up to 5 years after treatment
  Acute and late toxicities evaluated according to the CTCAE v5.0 classification :
  1. Acute toxicity is defined as toxicity observed between the start of RT and up to 3 months after the end of RT.
  2. Late toxicity is defined as toxicity observed between 3 months and 5 years after the end of radiotherapy.
  3. Late toxicity will be evaluated at 3 and 5 years.
Quality of life evaluation | Up to 5 years after treatment
  Quality of life evaluated by the EORTC QLQ-C30 questionnaire at each consultation (initial, end of radiotherapy, and at each follow-up (every 3 months after treatment)
Evaluation of the evolution of the tumour marker CA 19.9 | Until the end of the follow-up
  Change in tumour marker CA 19.9 from baseline to follow-up
Dosimetric benefits of daily adaptation, for each dosimetric parameter (GTV and PTV coverage, organs at risk doses), by comparing the average results obtained for each patient over all sessions with the 'adapted' plan compared to the 'predicted plan' | At the end of the treatment
  Collection of the dosimetric results obtained in terms of dose/volume on the projected dosimetry (coverage of the PTV by the prescription dose on the total dosimetry, dose received at GTV....) ; Collection and summation of dosimetric results obtained in terms of dose/volume for adaptive radiotherapy sessions and comparison with predictive dosimetry
Correlation between dosimetry and outcomes (local control, toxicities) | At the end of the treatment
  Correlation of PTV coverage and GTV dose with local control, progression-free survival and overall survival (predictive and adaptive dosimetry) ; Correlation of the dose received in organs at risk (duodenum, small intestine, stomach, colon) with the occurrence of acute and late digestive toxicities (predictive and adaptive dosimetry)

CONTACTS AND LOCATIONS:
Locations (17):
- France (17):
  - Centre d'Oncologie du Pays-Basque, Bayonne
  - Institut Bergonié, Bordeaux
  - CHU Brest, Brest
  - Centre Hospitalier Carcassone, Carcassonne
  - Centre Jean PERRIN, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Institut Paoli-Calmettes, Marseille
  - Institut régional du Cancer de Montpellier, Montpellier
  - CHU Nîmes, Nîmes
  - Hôpital européen Georges-Pompidou, Paris
  - Hôpital Tenon AP-HP, Paris
  - HU Pitié-Salpêtrière, Paris
  - CHU Bordeaux Haut-Lévêque, Pessac
  - Centre Eugène Marquis, Rennes
  - Institut Claudius Regaud, Toulouse
  - ORLAM, Villeurbanne

IPD SHARING:
Plan to Share IPD: No